CLINICAL TRIAL: NCT04230863
Title: Neuroplasticity-Based Cognitive Remediation for Chemotherapy-Related Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: University of Utah (Other)
Responsible Party: Principal Investigator, Paul Newhouse, MD, Principal Investigator, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 191394
Record Dates: First submitted 2020-01-10; First posted 2020-01-18 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Cancer Survivors; Chemotherapy-related Cognitive Impairment
Keywords: Chemotherapy; Cognitive Impairment; neuroplasticity-based computerized cognitive remediation; nCCR
MeSH Terms: conditions — Chemotherapy-Related Cognitive Impairment; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: A single-arm, open label design; All analyses are pre-post, with participants serving as their own controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neuroplasticity-based Computerized Cognitive Remediation (Experimental): Participants will receive a 45-hour of Neuroplasticity-based Computerized Cognitive Remediation.
  Interventions: Behavioral: Neuroplasticity-based Computerized Cognitive Remediation

INTERVENTIONS:
Behavioral: Neuroplasticity-based Computerized Cognitive Remediation — The nCCR has two major components: Bottom up and Top down training. "Bottom up" training: The training includes selected tasks from "Brain HQ", a program designed for older adults, that enhances basic processing of sensory stimuli with the goal to improve fidelity of auditory and visual encoding.
  "Top down training": We designed programs to target cognitive control functions associated with poor treatment response, i.e., initiation and use of verbal strategy and susceptibility to interference. These "Top Down" Programs include a visual attention program, either Catch the Ball or Neurogrow, and a semantic strategy program, Semantic Organization.

SUMMARY:
The investigators propose to apply neuroplasticity-based computerized cognitive remediation (nCCR) to treat chemotherapy-related cognitive impairment (CRCI).

DETAILED DESCRIPTION:
Advances in cancer treatment are producing a growing number of cancer survivors; therefore, issues surrounding quality of life during and following cancer treatment have become increasingly important. Chemotherapy-related cognitive impairment (CRCI) is one such quality of life issue that is commonly reported following chemotherapy treatment in adults. Although studies reporting cognitive impairments associated with chemotherapy have been reported since the 1980s, the phenomenon commonly referred to as 'chemo brain' or 'chemo fog' is poorly understood, and for some patients becomes the most distressful survivorship issue faced. Studies suggest that while up to up to 75% exhibit cognitive decline during treatment, many patients will return to their pre-chemo level of functioning 1 year after completing treatment. However, for 30-35% of cancer patients, their cognitive issues persist.

Studies suggest that this persistent chemotherapy-related cognitive impairment (pCRCI) can remain for months to years after completing treatment, which may have implications for the trajectory of how both normal cognitive aging occurs, but also the risk of cognitive disorders such as Alzheimer's disease, for the growing number of long-term cancer survivors. These concerns are particularly relevant for older individuals as risk for not only cancer, but cognitive impairment (such as dementia) increases with age. As of January 2016, 62% of cancer survivors (9.61 million) are currently 65 years or older, and this number is expected to increase dramatically over the coming decades. Therefore, as the number of older cancer survivors who have will have to cope with pCRCI is likely to increase, it is crucial that The investigators understand the cognitive impairments, the impact on survivors' functioning, and develop treatments for pCRCI.

The investigators propose to target cognitive deficit in CRCI using a novel cognitive enhancement strategy. Our choice of cognitive focus is informed by clinical, behavioral and neurobiological data suggesting a reliable association between cognitive control deficits (CCD), damage to the cognitive control network (CCN), and decline in cognitive functioning. The CCN is a neural network that supports important cognitive control functions such as alerting and orienting attention, response selection, cognitive flexibility, strategy generation, and inhibition of prepotent responses. The investigators propose to apply neuroplasticity-based computerized cognitive remediation (nCCR) to the treatment of CRCI as it has demonstrated training and transfer effects of enhanced CCN function in a similar, abnormally aging population. The theory guiding neuroplasticity-based cognitive interventions is that network abnormalities associated with negative disease-specific clinical outcomes can be altered through the induction of neuroplasticity (even in the aging brain) resulting in enhanced functioning of the target network, and symptomatic improvements.

ELIGIBILITY:
1. Inclusion Criteria:

   All participants will:
   1. Be between 35 and 80 years of age,
   2. Have been diagnosed with noninvasive or invasive (Stage 1, 2, or 3A) breast cancer, colon cancer, lymphoma, endometrial cancer or ovarian cancer
   3. Have undergone treatment with systemic chemotherapy within the last 1-8 years,
   4. Endorse persistent CRCI subjective complaints (as defined below),
   5. Have no active cardiac, neurologic, or psychiatric illness,
   6. Fluent in and able to read English.
2. Exclusion Criteria:

Participants will be excluded for:

1. Any active neurologic psychiatric disease, clinically significant cognitive impairment or dementia, history of significant head trauma followed by persistent neurologic deficits, or known structural brain abnormalities,
2. Current major depression or another major psychiatric disorder as described in DSM-5 (use of CNS active medications (e.g. antidepressants) will be permitted, provided dosing has been stable for at least 3 months),
3. Any history of alcohol or substance abuse or dependence within the past 2 years (DSM-5 criteria),
4. Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol.
5. Use of any investigational drugs within 30 days or 5 half-lives, whichever is longer, prior to screening, and
6. Use of cholinergic agents will be discouraged but will be reviewed on a case-by-case basis by the PI.
7. Red-green color blindness. Other types of color blindness will be reviewed on a case-by-case basis by the PI.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluate completion rates of nCCR | 2 years
  Assess the percentage of enrolled participants who completed of the 40-hour nCCR treatment
Evaluate visit frequency throughout nCCR treatment | through study completion, an average of 5 weeks.
  Assess the frequency of visits during nCCR treatment
Evaluate visit duration throughout nCCR treatment | through study completion, an average of 5 weeks.
  Assess the duration of visits during nCCR treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Newhouse, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No